CLINICAL TRIAL: NCT04805372
Title: Application of the Training Bundle With Video Demonstration and Video Feedback as the Core in the Teaching of Right Internal Jugular Vein Catheterization Skills
Brief Title: Video Demonstration and Video Feedback to Reduce Time to Perform Central Vein Cannulation in Junior Residents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021-0083
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Venous Puncture; Students, Medical; Education, Medical
Keywords: medical skill training; video modeling; video feedback; venous puncture; phlebotomy; medical education

STUDY DESIGN:
Intervention Model Description: Before the allocation, the instructor led the trainees to watch the demonstration video of the central vein operation and explained the main points of the operation at least 5 times.Before the operation, trainees should complete the operation-related test questions. And trainees should complete at least one central venipuncture model training and one actual operation under the personal guidance of the instructor before allocation.They will then be assigned to review a video of an expert performing central vein operation (VD alone), or both the expert video and a video of their own most recent operation(VD+VF), before returning to do another central vein operation. This will be repeated for a total of 5 central vein operation encounters and 5 video reviews.In the second week, each trainee completed at least 5 independent operations under the supervision of the instructor.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Students and teachers are not blinded, but researchers and data evaluators are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VD+VF group (Experimental): where they should review a video of an expert performing central vein operation and a video of their own most recent operation, before returning to do another operation. This will be repeated for a total of 5 central vein cannulation encounters and 5 video reviews.
  Interventions: Other: VD+VF group
- VD group (Placebo Comparator): where they should review a video of an expert performing central vein operation before returning to do another operation. This will be repeated for a total of 5 central vein cannulation encounters and 5 video reviews.
  Interventions: Other: VD group

INTERVENTIONS:
Other: VD+VF group — where they should review a video of an expert performing central vein operation and a video of their own most recent operation, before returning to do another operation. This will be repeated for a total of 5 central vein cannulation encounters and 5 video reviews.
  Arms: VD+VF group
Other: VD group — where they should review a video of an expert performing central vein operation before returning to do another operation. This will be repeated for a total of 5 central vein cannulation encounters and 5 video reviews.
  Arms: VD group

SUMMARY:
Central venous catheterization technique is a compulsory clinical skill for anesthesia resident physician. Because it is difficult to operate and may cause serious complications, teaching this skill is a key and difficult point in clinical teaching of anesthesiology department.This project aims to observe the effect of video demonstration combined with video feedback teaching on the central venous catheterization time of junior residents and to obtain a better training method for central venous catheterization skills.

DETAILED DESCRIPTION:
Central venous catheterization technology is a compulsory clinical skill for resident physicians. Because of its difficulty in operation and the possibility of serious complications, teaching this skill is a key and difficult point in clinical teaching in anesthesiology. This skill training has gone through the traditional "apprentice mode" teaching to the current video demonstration teaching, bedside feedback teaching, etc.. The attempts of multiple teaching modes are to help low-age resident doctors master the technology as soon as possible, improve the operation success rate, and reduce the incidence of complications.

The Department of Anesthesiology in our hospital is a key base for the standardized training of anesthesiologists in China. In recent years, the introduction of video demonstration methods for the central venous catheterization technology of low-age residents has achieved some results. Residents watch the demonstration operation videos specially recorded by the department, and perform operation exercises after passing the pre-operation assessment. The trainees self-reported that the teaching mode increased their confidence in learning this skill. However,in the actual training process, bedside comments (feedback teaching) were also involved, and it was discovered that it could cause panic and dissatisfaction of the patient, which was later improved into the paper-based feedback of the teacher.

The video demonstration teaching method was first applied to athletes' competitive training and was found to be effective in improving athletes' competitive skills.It was also used in medical education for surgical operation training, such as laparoscopic operation, which also obtained significant results. Feedback, as a method of attracting learners, has long been regarded as an important part of learning in medical education. We used bedside feedback teaching in the early stage, which was criticized by patients. Research has shown that video feedback may not only be superior to traditional verbal feedback methods alone, but it can also avoid problems from patients. When learners watch their own operation videos, video feedback will occur regardless of whether there is guidance from the instructor. Learners can watch these videos individually or with the teacher who can provide guidance at the same time. This teaching method is believed to be helpful for the assessment of skills. The use of video feedback originated from track and field sports learning. A large number of studies have found that video feedback teaching can be used as an effective means of medical communication skills training. Recently, it has also be used in clinical skills teaching. Current studies have confirmed that this teaching method can improve students' confidence in learning skills, but there is still relatively little research on skill acquisition.

In summary, video demonstration teaching and video feedback teaching are both useful in deliberate practice teaching (such as skill operation training). Skills operation training involves targeted repetitive exercises to improve skills, and feedback is the key to strengthening clinical learning. By video demonstrations, learners can observe and analyze the performance of experts (demonstrators) at key decision points under the guidance of the teacher. And video feedback can help promote self-assessment. It shows that the combination of the two may be more conducive to the integration of observational learning, imitation and self-evaluation, and speed up the progress of skill training. This joint teaching has been studied in sports research, while there are few studies in medical education. At present, a small study found that compared with oral feedback, the combined method can achieve better hernia repair skills, and there are recent research reports in peripheral vein indwelling operation training. But whether it is also suitable for the operation training of high-risk skills with greater difficulty coefficient, it needs to be confirmed by further research.

This project intends to observe the impact of video demonstration combined with video feedback teaching on the central venous catheterization time of low-age resident physicians, aiming to obtain a better method of central venous catheterization skills training, and to improve the learning confidence of students to better master this skill, improve the success rate of operation, reduce complications, and promote the application.

ELIGIBILITY:
Inclusion Criteria:

* The target population will be junior residents of the Department of Anesthesiology, the Second Affiliated Hospital of Zhejiang University with < 3 previous encounters performing central vein operation

Exclusion Criteria:

* The target population will be junior residents of the Department of Anesthesiology, the Second Affiliated Hospital of Zhejiang University with ≥ 3 previous encounters performing central vein operation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Average time required to complete 5 independent operations in the second week | in the second week
  In the second week, 5 operations were completed under the supervision of the instructor and the required time was recorded

SECONDARY OUTCOMES:
The puncture success rate and complications in the first week | in the first week
  The success and complications of each puncture were recorded
The puncture success rate and complications in the second week | in the second week
  The success and complications of each puncture were recorded
Training satisfaction of trainees | the day after the training
  After the training, questionnaire was used to survey the trainees' satisfaction with the training
Operation success rate and complications in 1 month after the training. | One month after the training
  Record the success rate and complications of each independent operation of the trainees after the end of the training
Operation success rate and complications in 3 month after the training. | One months after the training
  Record the success rate and complications of each independent operation of the trainees after the end of the training

CONTACTS AND LOCATIONS:
Overall Officials: lina Yu, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No